CLINICAL TRIAL: NCT01393028
Title: Computed Tomography Versus Exercise Testing in Suspected Coronary Artery Disease
Acronym: CRESCENT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Koen Nieman, Dr K Nieman, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRESCENT-11
Record Dates: First submitted 2011-06-27; First posted 2011-07-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Angina Pectoris; Chest Pain
Keywords: coronary artery disease; angina pectoris; Stable chest pain complaints
MeSH Terms: conditions — Angina Pectoris; Chest Pain; Coronary Artery Disease | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardiac CT (Experimental): Cardiac CT (CT calcium and/or CT angiography), followed by stress testing, invasive angiography or neither depending on the CT scan result
  Interventions: Other: Cardiac CT
- Standard care (Other): Standard diagnostic management, including stress testing and/or invasive angiography
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Cardiac CT — Cardiac CT: calcium scan and CT coronary angiography
  Arms: Cardiac CT
Other: Standard care — Standard care according to international guidelines
  Arms: Standard care

SUMMARY:
Direct non-invasive coronary imaging by computed tomography (CT) has the potential to improve the workup of patients with stable chest pain complaints. The objective of the study is to compare in a randomized fashion the effectiveness and efficiency of a CT angiographic driven workup of suspected coronary artery disease in comparison to the standard workup using stress testing.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years.
* Stable symptoms of chest pain or dyspnea potentially caused by obstructive CAD.

Exclusion Criteria:

* A history of surgical or percutaneous coronary revascularization
* Non-revascularized angiographic obstructive coronary artery disease (>50% diameter reduction).
* Normal invasive coronary angiography or stress imaging less than 1 years ago.
* Inability or unwillingness to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2011-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Chest pain | 1 year
  Reduction of chest pain symptoms by standardized questionnaire, at one year follow-up
Class IA Revascularizations | 1 year
  Number of revascularizations with an ESC class 1A indication

SECONDARY OUTCOMES:
Overall medical expenses | 1 year
  Overall medical expenses
Cost-effectiveness | 1 year
  Cost-effectiveness analysis based on the overall quality of life and medical expenses at one year.
Radiation dose | 1 year
  Cumulative radiation exposure at one year
Major adverse cardiovascular events | 1 year
  Composite endpoint of adverse cardiovascular events, including:
  All-cause mortality Non-fatal myocardial infarction Unstable angina requiring hospital admission Late revascularization procedures (>6 months after initial evaluation)
Quality of life | 1 year
  Change of quality of life at 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - MC Haaglanden, Leidschendam
  - Erasmus MC, Rotterdam
  - Havenziekenhuis, Rotterdam
  - Maasstadziekenhuis, Rotterdam

REFERENCES:
- [Derived] Lubbers M, Coenen A, Bruning T, Galema T, Akkerhuis J, Krenning B, Musters P, Ouhlous M, Liem A, Niezen A, Dedic A, van Domburg R, Hunink M, Nieman K. Sex Differences in the Performance of Cardiac Computed Tomography Compared With Functional Testing in Evaluating Stable Chest Pain: Subanalysis of the Multicenter, Randomized CRESCENT Trial (Calcium Imaging and Selective CT Angiography in Comparison to Functional Testing for Suspected Coronary Artery Disease). Circ Cardiovasc Imaging. 2017 Feb;10(2):e005295. doi: 10.1161/CIRCIMAGING.116.005295. PMID 28174196